CLINICAL TRIAL: NCT06672003
Title: Assessment of the Prevelance of Chronic Pain and Its Relationship to Frailty in Older Adults
Brief Title: Assessing the Relationship Between Chronic Pain and Frailty in Older Adults
Status: Completed | Type: Observational
Sponsor: Celal Bayar University (Other)
Responsible Party: Sponsor
Other Study IDs: MCBU-SM-FM-01
Record Dates: First submitted 2024-08-09; First posted 2024-11-04 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Chronic Pain; Frailty
MeSH Terms: conditions — Chronic Pain; Frailty | interventions — Hand Strength

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: 4 meter walking speed and hand grip strength — 4 meter walking seconds are noteed for each of participants

SUMMARY:
Pain is an unpleasant emotional sensation related to one's past experiences, originating from a certain part of the body, due to tissue damage or not. Pain is the most commonly reported symptom in the elderly. Chronic pain is persistent or recurrent pain lasting more than 3 months. It is a maladaptive process or a disease that requires multimodal treatment that causes functional decline, independent of the healing process, accompanied by affective, cognitive and motivational disorders, and deterioration in quality of life. Frailty: It is defined as a clinical condition characterized by weakness, physical disability, functional regression, inadequacy in activities of daily living, and increased dependence, which develops as a result of the decrease in physiological reserves in the body with age. It has been reported that the risk of falls, disability, hospitalization and premature death is higher in the frail elderly. The prevalence of vulnerability in societies varies. Frailty rates ranging from 4 to 59% have been reported in developed and developing countries. In this study, it was aimed to evaluate whether there is a relationship between chronic pain and frailty in individuals aged 65 and over.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic pain who are registered with a family medicine unit

Exclusion Criteria:

* Having an active malignancy,
* having a physical disability,
* being bedridden,
* having a psychotic disorder,
* having a cognitive disorder, and refusing to participate.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: The universe of the study consists of all individuals aged 65 and over registered in a family health center. Participants to be included in the study from this universe will be determined using the stratified random sampling method.
Sampling Method: Probability Sample
Enrollment: 203 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
frailty | 12 months
  Participants' frailty levels will be determined.
chronic pain | 6 months
  The relationship between participants' frailty levels and chronic pain frequency will be examined.

CONTACTS AND LOCATIONS:
Locations (1):
- Manisa Celal Bayar University, Manisa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
upon request of the board

DOCUMENTS (1):
  • Study Protocol (2024-08-16): https://cdn.clinicaltrials.gov/large-docs/03/NCT06672003/Prot_000.pdf